CLINICAL TRIAL: NCT05290324
Title: Propofol or Midazolam for Sedation and Early Extubation Following Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chaudhry Pervaiz Elahi Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, Shumaila rai, Principal Investigator, Chaudhry Pervaiz Elahi Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPEIC22
Record Dates: First submitted 2022-01-30; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass graft; midazolam; propofol
MeSH Terms: conditions — Coronary Artery Disease | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Radomized Controlled Trial
Who Masked: Participant
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIdazolam Group (Experimental): Following surgery Immediately after shifting in ICU, midazolam infusion were administered as 0.25 mg/kg/min.
  Interventions: Drug: Midazolam
- Propofol Group (No Intervention): Following surgery after Immediately shifting in ICU propofol infusion was started at 10µg/kg/min.

INTERVENTIONS:
Drug: Midazolam — Midazolam infusion will be given after the surgery as 0.25 mg/kg/min.
  Other Names: Versed
  Arms: MIdazolam Group

SUMMARY:
Propofol and midazolam are used frequently as sedating agents among patients who undergo coronary artery bypass graft surgery but no study in Pakistan has been done to compare their effectiveness aiming early extubation.

DETAILED DESCRIPTION:
Propofol is an intra lipid and alkali phenol chemically it is unrelated to sedative agents or anaesthetic. Midazolam is a banzodiazepen. Most of its properties are similar to diazepam. It is a common practice to use sedatives to provide comfort and decrease "ventilator-asynchrony" in critically ill patients that may require prolonged invasive mechanical ventilation. The other reason to employ sedatives is to reduce the anxiety associated with the inaviseve procedures routinely conducted in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) III who were selected for coronary artery bypass graft surgery.

Exclusion Criteria:

* History of any psychiatric disease.
* Using antidepressants
* Alcohol abusers
* Obese
* Pregnant women

Ages: 20 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Duration of post-surgery sedation | Time in minutes calculated from end of surgery to the time of awakening up to 24 hours in both study groups
  Duration of post-surgery sedation following cardiac surgery
Time taken to post-surgery extubation | Time taken in minutes from the end of the cardiac surgery to post-surgery extubation up to 1 week duration in both study groups
  Time taken from the end of cardiac surgery to post-surgery extubation

CONTACTS AND LOCATIONS:
Overall Officials: Shumaila Rai, MBBS, Principal Investigator — Ch. Pervaiz Elahi Institute of Cardiology, Multan, Pakisan
Locations (1):
- Ch. Pervaiz Elahi Institute of Cardiology, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No